CLINICAL TRIAL: NCT06166173
Title: Using Color Doppler US Artifact to Identify Localization of Breast and Axilla Tumor Markers
Brief Title: Using Color Doppler US Artifact to Identify Tumor Markers
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Murat Asik, Assistant professor, Istanbul Medeniyet University
Other Study IDs: BREAST TM
Record Dates: First submitted 2023-11-24; First posted 2023-12-12 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Breast Cancer; Interventional Radiology; Doppler Ultrasound
Keywords: breast cancer; tumor marker; doppler ultrasound; neoadjuvan chemotherapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Breast tumor: Female patients with breast tumors and/or axillary lymph node metastases who had markers placed before neoadjuvant chemotherapy (NACT), and patients undergoing preoperative marker localization after NACT

SUMMARY:
Before neoadjuvant chemotherapy (NACT) in cases of locally advanced breast cancer, malignant masses in the breast and biopsy-proven tumor involvement axillary lymph nodes are marked with metallic markers. The primary objective of this marking is to establish the precise localization of the tumor which response to NACT partial or completely. However, selecting the marker with ultrasound (US) proves challenging in many instances. Research studies indicate that patients with occult markers are observed at a frequency of 24%. Some studies propose that the twinkling artifact serves as a reliable method for accurately indicating the localization of certain tumor markers. This artifact is deemed particularly helpful for lesions situated in the axilla or posterior of the breast, which may not be visible with US and are undetectable with mammography.

In the context of Color Doppler examination, the investigators have noted the presence of another color Doppler artifact which can aid in determining marker localization. When the pulse repetition frequency (PRF) is reduced and the color gain is increased, color noise, termed as color confusion or blooming artifact/effect, is observed within the color steer. While this color confusion tends to mask healthy tissues, it has been observed that the tumor marker remains unaffected by the blooming effect. Consequently, this artifact serves to distinctly reveal the borders and localization of the tumor marker.

In some studies, it has been stated that the twinkling artifact, which is a color Doppler artifact and whose mechanism is not fully understood, is a reliable method to accurately indicate the localization of some tumor markers. It has been reported that this artifact will be very helpful, especially in lesions located in the axilla or posterior of the breast, which cannot be seen with US and cannot be detected with mammography .

In Color Doppler examination, we saw that another color Doppler artifact, such as the twinkling artifact, could also be helpful in determining marker localization. When the PRF is reduced and the color gain is increased, color noise, which is selected as color confusion and can be called blooming artifact or blooming effect-like, is observed in all structures within the color steer. While healthy tissues are masked by this color confusion, the tumor marker is protected from the blooming effect. Thus, with this artifact, tumor marker borders and localization are clearly revealed.

DETAILED DESCRIPTION:
Following an exhaustive review of the existing literature, the investigators have determined that their study stands as the first to show the utility of like blooming artifact appearance in color Doppler US for precisely determining the localization of tumor markers placed in the breast and axilla. There are two crucial phases in this study: Pre and post-NACT patients. In these two stages, tumor markers could be successfully demonstrated using this artifact (blooming artifact-like appearance). This groundbreaking finding lends support to B-mode ultrasound (US), which demonstrates high diagnostic potential and proves valuable for radiologists, thereby providing reassurance Post-NACT, the hypoechoic mass in the breast and the thick-cortical lymph node in the axilla undergo shrinkage. Identifying the residual mass becomes feasible solely with the hyperechoic marker placed before NACT. The hyperechoic marker in the shrinking mass after NACT cannot be discerned from the hyperechoic fibrous structures in the normal breast parenchyma. However, when the like blooming artifact is generated in the color Doppler examination, the echogenic normal breast or axillary parenchyma is enveloped by this artifact. Importantly, the metallic marker remains unaffected by this artifact.

To achieve homogeneity of this artifact, specific Doppler US parameters must be applied to the color Doppler examination window. For this artifact to be diagnostic, color Doppler US must be provided in the all examination consistently. Consequently, while the non-marker area is covered with the blooming artifact, the marker becomes distinctly visible.

The investigators note that while the use of twinkling artifacts in determining marker localization is well-established, the blooming artifact utilized in this study remains unknown. No prior literature research has explored this artifact or highlighted its diagnostic contributions.

In this study, the investigators have aimed to mask tissues outside the marker with the blooming artifact. Consequently, the linear marker cannot be masked and appears echogenic. In the color Doppler US window covered with the blooming artifact, only the marker itself stands out as a smooth linear echogenicity. This distinctive feature enables an easy examination for determining marker localization, irrespective of the marker's structure, shape, or ambient temperature. Therefore, it can be asserted that this method is not only easier to implement but also more reliable compared to other techniques.

ELIGIBILITY:
Inclusion Criteria:

* patients who have breast cancer and will receive NACT,
* patients who are scheduled for breast-conserving surgery,
* those who are not allergic to metals

Exclusion Criteria:

* patients with breast cancer for whom NACT is not planned,
* patients with bleeding disorders, patients with metallic allergies,
* patients with cooperation problems and those who cannot remain still during US

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with breast cancer and/or pathologically proven axillary lymph node involvement and who are planned or have received NACT
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Easier localization of breast tumor marker with Doppler ultrasound findings in approximately 20 patients | through study completion, an average of 6 months
  Use of Doppler US artifacts as an auxiliary diagnostic method in cases where tumor markers in the breast and axilla cannot be detected with conventional US.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medeniyet University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/37326508/